CLINICAL TRIAL: NCT01046942
Title: ThrombElastoGraphic Haemostatic Status and Antiplatelet Therapy After Coronary Artery Bypass Graft Surgery(TEG-CABG Trial):Does Intensified Postoperative Antiplatelet Therapy in Preoperatively Identified Hypercoagulable Patients Improve Outcome After CABG Surgery
Brief Title: ThrombElastoGraphic Haemostatic Status and Antiplatelet Therapy After Coronary Artery Bypass Graft Surgery
Acronym: TEG-CABG
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Sulman Rafiq, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-C-2007-0057
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2013-09-24 (Estimated); Status verified 2013-09

CONDITIONS: Graft Patency; Coronary Artery Bypass Grafting Surgery; Hypercoagulability; Thrombosis
Keywords: Saphenous vein; Antiplatelet therapy; Hypercoagulable; Clopidogrel resistance; Aspirin resistance; Clopidogrel; Aspirin; Saphenous vein graft disease; TEG; Thrombelastography; Multiplate aggregometry; Multislice CT; Coronary artery bypass graft surgery; coagulation status; graft patency; CABG
MeSH Terms: conditions — Thrombophilia; Thrombosis | interventions — Clopidogrel; Aspirin; aspirin, magnesium oxide combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clopidogrel+Aspirin, hypercoagulabel (Experimental)
  Interventions: Drug: Clopidogrel+acetylsalicylic acid
- Aspirin,hypercoagulabel control (Active Comparator)
  Interventions: Drug: acetylsalicylic acid

INTERVENTIONS:
Drug: Clopidogrel+acetylsalicylic acid — loading dose clopidogrel 300mg on second postoperative day. Thereafter 75mg clopidogrel daily for 3 months Aspirin 75mg daily, started within 24 hours after surgery
  Other Names: Plavix
  Arms: Clopidogrel+Aspirin, hypercoagulabel
Drug: acetylsalicylic acid — aspirin 75 mg daily, started 6-24 hours after surgery
  Other Names: Aspirin; Magnyl
  Arms: Aspirin,hypercoagulabel control

SUMMARY:
The purpose of this study is to determine whether adding clopidogrel to aspirin after coronary bypass operation (CABG) improves graft patency, in patients that have preoperatively increased platelet activity(hypercoagulable) and therefore greater risk of graft occlusion( thrombosis).

DETAILED DESCRIPTION:
Graft patency after CABG is reported to 80-90% worldwide 1 year following surgery. In the immediate period after surgery, and the following month, graft occlusion mainly occurs due to thrombosis.

Patients with platelet hyperreactivity have increased risk of thromboembolic events, including graft occlusion, myocardial infarction and stroke. Therefore intensifying the antiplatelet therapy in these patients, must be anticipated to have beneficial effects.

Hypercoagulable patients are identified with thrombelastography(TEG) as having a Maximal Amplitude(MA)>69, thereafter randomized to either clopidogrel(3months) and aspirin or aspirin alone. At 3 months postoperative after surgery the coronary graft patency is assessed with Multislice CT scan.

Pre- and postoperatively, and then again at 3month followup, TEG and multiplate aggregometry are performed to assess platelet reactivity and resistance to aspirin and clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Elective/subacute multivessel CABG
* Isolated CABG procedure, no concomitant surgery
* age > 18 years
* Able to give informed consent

Exclusion Criteria:

* Myocardial infarction <48h of surgery
* Prior CABG surgery within 1 month
* Cardiac Shock within 48h of surgery
* Atrial fibrillation
* Anticoagulation therapy with VKA
* ICH/TCI within 30 days
* Prior peptic ulcer· Platelet count < 150 E9
* Ongoing bleeding
* Known platelet disease
* Allergic to aspirin or clopidogrel
* Liver disease with elevated ALAT/ASAT> 1,5x normal
* Creatinine> 0,120mmol/l
* Contrast allergy
* Alcohol or narcotics abuse
* Pregnancy
* Not able to give informed consent
* Geographically not available for follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2008-11; Primary Completion 2014-05 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Graft patency at 3 months | 3 months
  Graft patency of Saphenous vein grafts will be significantly higher in TEG-Hypercoagulable patients on clopidogrel+aspirin vs. aspirin alone.

SECONDARY OUTCOMES:
Rate of other thromboembolic events( e.g. myocardial infarction,stroke, pulmonary embolus etc.)and cardiovascular death | 3 months
  In the TEG-Hypercoagulable intervention group (clopidogrel+aspirin) we expect significantly lower rates, of other thromboembolic events (e.g. myocardial infarction,stroke, pulmonary embolism etc) and cardiovascular death, compared to TEG-Hypercoagulable patients on aspirin monotherapy.
Assessing coagulation profile pre- and postoperatively, including aspirin and clopidogrel resistance | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sulman Rafiq, MD, Study Director — Dept. of Cardiothoracic Surgery, Rigshospitalet, Copenhagen University Hospital; Daniel Steinbrüchel, Professor, Principal Investigator — Dept. of Cardiothoracic Surgery, Rigshospitalet, Copenhagen University Hospital; Pär Johansson, cons. MD,MPA, Study Director — Blood Bank, Rigshospitalet, Copenhagen University Hospital; Klaus Kofoed, cons.MD, Study Chair — Dep. of Cardiology, Rigshospitalet,Copenhagen University Hospital; Mette Zacho, MD, Study Chair — Dept. of Radiology, Rigshospitalet, Copenhagen University Hospital; Trine Stissing, MD, Study Chair — Blood Bank, Rigshospitalet, Copenhagen University Hospital
Locations (1):
- Dep. of cardiothoracic surgery, Rigshospitalet, Copenhagen, Kbh, Denmark

REFERENCES:
- [Derived] Rafiq S, Johansson PI, Zacho M, Stissing T, Kofoed K, Lilleor NB, Steinbruchel DA. Thrombelastographic haemostatic status and antiplatelet therapy after coronary artery bypass surgery (TEG-CABG trial): assessing and monitoring the antithrombotic effect of clopidogrel and aspirin versus aspirin alone in hypercoagulable patients: study protocol for a randomized controlled trial. Trials. 2012 Apr 27;13:48. doi: 10.1186/1745-6215-13-48. PMID 22540524